CLINICAL TRIAL: NCT06963749
Title: Pain Control During Brief Intervention in Deep Sedation: no Pain or no Memory
Brief Title: Surgical Intervention in Deep Sedation: No Pain or no Memory
Acronym: SedNOL
Status: Completed | Type: Observational
Sponsor: ASL Novara (Other Government)
Responsible Party: Principal Investigator, Davide Colombo, Director Anesthesia and Intensive Care Unit, ASL Novara
Other Study IDs: SedNol
Record Dates: First submitted 2024-08-08; First posted 2025-05-09 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-08

CONDITIONS: Pain, Acute; Surgical Procedure, Unspecified
Keywords: Deep sedation; Nociception; NOL index; Pain control
MeSH Terms: conditions — Acute Pain; Agnosia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study group: All patients meeting the inclusion criteria who underwent surgical brief procedures in deep sedation

SUMMARY:
The goal of this observational study is to assess the levels of nociception in deeply sedated patients who need painful and short-duration surgical procedure.

The main question it aims to answer is to verify that the sedative protocols used in clinical practice are sufficiently effective also in terms of nociception.

Participants will deeply sedated and monitored with PMD-200™ to detect the nociception level (NOL Index).

DETAILED DESCRIPTION:
Prior to enrollment, upon arrival in the operating room and after being properly positioned on the operating table, patients will undergo standard intraoperative monitoring with pulse oximetry (SpO2), 3-lead electrocardiography (ECG), non-invasive brachial blood pressure monitoring (BP), a sensor for the Bispectral Index (BIS), and a nociception sensor (NOL) will also be placed.

Patients will be pre-oxygenated with a face mask with inspired oxygen fraction (FiO2) at 100% for 3 minutes.

The induction phase of deep sedation anesthesia will be conducted with a single bolus of Fentanyl 1 mcg/kg and total intravenous anaesthesia - target controlled infusion (TIVA-TCI) Propofol with an effect site concentration (Cε) of 4.0 mcg/mL.

Once the sedation level shows a Bispectral Index between 40 and 60, observation of the NOL Index will begin.

Subsequently, the laryngeal mask can be positioned, mechanical ventilation started, and the surgical procedure commenced.

During this phase, the maintenance of the anesthetic plan will be ensured by the infusion of Propofol in TIVA-TCI (with a Cε that keeps the BIS between 40 and 60) and the administration of Paracetamol 1 g, Ketorolac 30 mg, and Dexamethasone 4 mg.

At the end of the surgical procedure, the observation of the NOL Index will conclude.

Upon awakening, patients will be taken to the Post-Anesthesia Care Unit (PACU), where they will remain until their vital parameters are stabilized. At this point, 15 minutes post-operatively, the intensity of pain will be recorded using the numeric pain rating scale (NRS) scale.

Subsequently, patients will be transferred to the ward, where, 2 hours post-operatively, they will be interviewed about the intensity of post-operative pain and whether they need any rescue analgesic doses.

Data collection and management will be handled by the investigator and/or the designated study staff.

Data will be collected directly into a digital file (spreadsheet - MS Excel - Microsoft, Redmond, CA) without the use of paper forms.

Data will be collected anonymously without identifying codes that could link to the patient's medical record and identity. The correspondence list between demographic data and the patients' identification codes will be kept at the enrolling center and will only be accessible to the study staff.

The data to be collected include the following:

1. Anthropometric Data:

   1. Sex
   2. Age
   3. Weight
   4. Height
   5. Body Mass Index (BMI)
   6. American Society of Anesthesiologists (ASA) Physical Status
2. Clinical Data

   1. Surgical Procedure Performed
   2. Heart Rate (HR)
   3. Non-Invasive Blood Pressure (BP)
   4. Pulse Oximetry (SpO2)
   5. Bispectral Index (BIS)
   6. NOL Index
   7. NRS Pain Scale

Continuous variables will be presented as mean and standard deviation or as median and interquartile range depending on their distribution. Normal distribution will be assessed using the Kolmogorov-Smirnov test. Any sub-analyses and comparisons between sub-groups will be conducted using the Student's t-test for parametric data, while the Mann-Whitney test will be used for non-parametric data. Categorical variables will be presented as absolute numbers and percentages of the total sample. Any sub-analyses and comparisons between sub-groups will be conducted using the Chi-square test or Fisher's exact test, depending on the size of the sub-groups. In all cases, the null hypothesis will be rejected for α values <0.05. The software used for data analysis and sample size calculation is MedCalc v. 22.013 (MedCalc Software, Ostend, Belgium).

ELIGIBILITY:
Inclusion Criteria:

* Adult patient
* ASA Physical Status I - II - III

Exclusion Criteria:

* ASA Physical Status IV
* Pregnant and breastfeeding patients
* Pre-existing cardiac arrhythmias
* Patients with neuromuscular diseases
* Patients with psychiatric syndromes under pharmacological treatment
* Patients with chronic use of analgesics
* Patients with a history of drug abuse
* Allergy to one or more drugs used in the protocol
* Refusal to consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population consists of patients from the Ss. Trinità Hospital in Borgomanero between March 1, 2024, and August 31, 2024, who are to undergo surgical procedures lasting less than 90 minutes and particularly painful, with an indication for deep sedation anesthesia.
Sampling Method: Non-Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2024-03-01 (Actual); Primary Completion 2025-01-31 (Actual); Study Completion 2025-01-31 (Actual)

PRIMARY OUTCOMES:
High level of nociception | The interval between reaching the appropriate level of sedation (Bispectral Index - BIS between 40 and 60) and the end of the surgical stimulation.
  The sedation protocol used will be considered ineffective in terms of nociception if the percentage of time during which the NOL index exceeds the threshold of 25, relative to the observation time, is greater than 25%.

SECONDARY OUTCOMES:
NOL Index >25 | The interval between reaching the appropriate level of sedation (Bispectral Index - BIS between 40 and 60) and the end of the surgical stimulation.
  Time in minutes during which the NOL index exceeds the threshold of 25
NOL Index Peaks | The interval between reaching the appropriate level of sedation (Bispectral Index - BIS between 40 and 60) and the end of the surgical stimulation.
  Number of peaks with a NOL index greater than 40

OTHER OUTCOMES:
Pain at 15th minute | 15th minute post-surgery
  Evaluate, if it exists, a correlation between the percentage of time during which the NOL index exceeds the threshold of 25 and the NRS scale at 15 minutes post-surgery.
Pain at 2nd hour | 2nd hour post-surgery
  Evaluate, if it exists, a correlation between the percentage of time during which the NOL index exceeds the threshold of 25 and the NRS scale 2 hours post-surgery.
Analgesic rescue | The interval between the end of the surgical stimulation and the 2nd hour post-surgery.
  Evaluate, if it exists, a correlation between the percentage of time during which the NOL index exceeds the threshold of 25 and the need for any rescue analgesic doses requested by the patient.

CONTACTS AND LOCATIONS:
Overall Officials: Davide Colombo, PhD, Study Director — ASL Novara
Locations (1):
- SS. Trinità Hospital, Borgomanero, Novara, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Coluzzi F. Intraoperative nociception: "if you can't measure it, you can't manage it". Minerva Anestesiol. 2019 May;85(5):462-464. doi: 10.23736/S0375-9393.19.13612-7. Epub 2019 Feb 13. No abstract available. PMID 30762333
- [Background] Ghanty I, Schraag S. The quantification and monitoring of intraoperative nociception levels in thoracic surgery: a review. J Thorac Dis. 2019 Sep;11(9):4059-4071. doi: 10.21037/jtd.2019.08.62. PMID 31656682
- [Background] Klein AA, Meek T, Allcock E, Cook TM, Mincher N, Morris C, Nimmo AF, Pandit JJ, Pawa A, Rodney G, Sheraton T, Young P. Recommendations for standards of monitoring during anaesthesia and recovery 2021: Guideline from the Association of Anaesthetists. Anaesthesia. 2021 Sep;76(9):1212-1223. doi: 10.1111/anae.15501. Epub 2021 May 20. PMID 34013531
- [Background] Meijer FS, Martini CH, Broens S, Boon M, Niesters M, Aarts L, Olofsen E, van Velzen M, Dahan A. Nociception-guided versus Standard Care during Remifentanil-Propofol Anesthesia: A Randomized Controlled Trial. Anesthesiology. 2019 May;130(5):745-755. doi: 10.1097/ALN.0000000000002634. PMID 30829658
- [Background] Meijer F, Honing M, Roor T, Toet S, Calis P, Olofsen E, Martini C, van Velzen M, Aarts L, Niesters M, Boon M, Dahan A. Reduced postoperative pain using Nociception Level-guided fentanyl dosing during sevoflurane anaesthesia: a randomised controlled trial. Br J Anaesth. 2020 Dec;125(6):1070-1078. doi: 10.1016/j.bja.2020.07.057. Epub 2020 Sep 17. PMID 32950246
- [Background] Won YJ, Lim BG, Lee SH, Park S, Kim H, Lee IO, Kong MH. Comparison of relative oxycodone consumption in surgical pleth index-guided analgesia versus conventional analgesia during sevoflurane anesthesia: A randomized controlled trial. Medicine (Baltimore). 2016 Aug;95(35):e4743. doi: 10.1097/MD.0000000000004743. PMID 27583920
- See also: Statement on Continuum of Depth of Sedation: Definition of General Anesthesia and Levels of Sedation/Analgesia — http://www.asahq.org/standards-and-practice-parameters/statement-on-continuum-of-depth-of-sedation-definition-of-general-anesthesia-and-levels-of-sedation-analgesia
- See also: General Anesthesia — http://www.issalute.it/index.php/la-salute-dalla-a-alla-z-menu/a/anestesia-generale

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-10-23): https://cdn.clinicaltrials.gov/large-docs/49/NCT06963749/Prot_SAP_001.pdf